CLINICAL TRIAL: NCT05807750
Title: Effects Of Income Supplements On 30-Day Readmissions For Vulnerable Older Adults: A Randomized, Controlled, 300-Subject Clinical Trial
Brief Title: Effects Of Income Supplements On 30-Day Readmissions For Vulnerable Older Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate eligible population size at recruitment site, resulting in inadequate pace of recruitment per funder guidance.
Sponsor: AltaMed Health Services Corporation (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-001 Sonik Readmit RCT; P30AG024968 (NIH)
Record Dates: First submitted 2023-03-23; First posted 2023-04-11 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Patient Readmission
Keywords: Patient Readmission; Income

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Enhanced care planning only (plus $15 as compensation for participation)
  Interventions: Other: Enhanced care planning
- Intervention (Experimental): Enhanced care planning plus a one-time $300 post-discharge income supplement
  Interventions: Other: Post-discharge income supplement; Other: Enhanced care planning

INTERVENTIONS:
Other: Post-discharge income supplement — $300 income supplement
  Arms: Intervention
Other: Enhanced care planning — Enhanced care planning provided by a nurse care manager

SUMMARY:
Unplanned 30-day hospital readmissions are an critical healthcare quality metric, with meaningful effects on patients and health systems operations. Interventions to reduce unplanned readmissions have primarily operated within a healthcare-centric frame, with enhancements to either pre- or post-discharge care planning, medication reconciliation, or visit frequency. Associations of 30-day readmission rates with poverty status and other social factors, however, suggest that attending to unmet social needs may yield added benefits to models focused on healthcare delivery. The purpose of the present trial is to provide evidence regarding the effects on 30-day readmissions of providing a one-time post-discharge income supplement to socially vulnerable older adults with medical complexity participating in an enhanced care coordination program.

ELIGIBILITY:
Inclusion Criteria:

* A participant in the underlying enhanced care planning program
* aged 55 years or older
* attending an outpatient clinic appointment as part of the underlying enhanced care planning program within 10 days of being discharged from an inpatient hospital stay
* able to understand the study consent form (with interpretation services if needed)

Exclusion Criteria:

* The candidate is not discharged from the index admission to a community setting (e.g., they will be excluded if they are discharged to a skilled nursing facility)
* The candidate has a legal guardian with control over financial decision-making
* The candidate has been approached about the study during a previous encounter
* The index hospitalization was a planned admission

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Unplanned 30-day readmission | Within 30 days of the index hospital discharge
  Whether a participant has an unplanned readmission within 30 days of the index hospital discharge

SECONDARY OUTCOMES:
30-day post-discharge medical expenditures | Within 30 days of the index hospital discharge
  Total medical expenditures in the 30 days after the index hospital discharge
90-day post-discharge medical expenditures | Within 90 days of the index hospital discharge
  Total medical expenditures in the 90 days after the index hospital discharge
30-day post-discharge medical readmission OR emergency department visit | Within 30 days of the index hospital discharge
  Whether a participant has an unplanned readmission OR emergency department visit within 30 days of the index hospital discharge
90-day post-discharge medical readmission OR emergency department visit | Within 90 days of the index hospital discharge
  Whether a participant has an unplanned readmission OR emergency department visit within 90 days of the index hospital discharge
Unplanned 90-day readmission | Within 90 days of the index hospital discharge
  Whether a participant has an unplanned readmission within 90 days of the index hospital discharge

OTHER OUTCOMES:
Post-discharge care plan adherence | Within 90 days of the index hospital discharge
  Clinic visit attendance, medication fills/refills

CONTACTS AND LOCATIONS:
Overall Officials: Rajan A Sonik, PhD, JD, MPH, Principal Investigator — Brandeis University
Locations (1):
- AltaMed Health Services Corporation, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calvillo-King L, Arnold D, Eubank KJ, Lo M, Yunyongying P, Stieglitz H, Halm EA. Impact of social factors on risk of readmission or mortality in pneumonia and heart failure: systematic review. J Gen Intern Med. 2013 Feb;28(2):269-82. doi: 10.1007/s11606-012-2235-x. Epub 2012 Oct 6. PMID 23054925